CLINICAL TRIAL: NCT00455507
Title: Placebo-controlled, Double-blind, Parallel Group, Fixed Dose Study of KW-6002 (Istradefylline) in the Treatment of Parkinson's Disease (Phase 2 Study)
Brief Title: A Phase 2b Study of Istradefylline (KW-6002) for the Treatment of Parkinson's Disease in Patients Taking Levodopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6002-0608
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 20 mg KW-6002 per day (two 10 mg tablets orally once daily for 12 weeks)
  Interventions: Drug: Istradefylline
- 2 (Experimental): 40mg KW-6002 per day (two 20 mg KW-6002 tablets orally once daily for 12 weeks)
  Interventions: Drug: Istradefylline
- 3 (Placebo Comparator): Two placebo tablets once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istradefylline — Two 10 mg KW-6002 tablets orally once daily for 12 weeks
  Other Names: KW-6002
  Arms: 1
Drug: Istradefylline — Two 20 mg tablets orally once a day for 12 weeks
  Other Names: KW-6002
  Arms: 2
Drug: Placebo — Two placebo tablets orally once daily for 12 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to establish the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the mean total hours of awake time per day spent in the OFF state in patients with advanced Parkinson's disease (PD) treated with levodopa.

DETAILED DESCRIPTION:
To establish the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the mean total hours of awake time per day spent in the OFF state in patients with advanced Parkinson's disease (PD) treated with levodopa. Patients who meet entry criteria will be randomized in a 1:1:1 ratio to double blind treatment with oral doses of 20 or 40mg/day istradefylline or matching placebo. Patients will be treated for 12 weeks and will have interim visits and end of treatment visit to assess the efficacy and safety of istradefylline.

ELIGIBILITY:
Inclusion Criteria:

1. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD.
2. PD stages 2-4 in the OFF state for Modified Hoehn and Yahr Scale.
3. On levodopa/dopa-decarboxylase inhibitor for at least one year.
4. Taking at least three doses and >=300mg of levodopa per day for at least four weeks before randomization.
5. Predictable end of dose wearing off.
6. Able to satisfactorily complete Hauser based 24-hour patient Parkinson's diary.
7. Have an average of two hours of OFF time on 24-hour diaries.
8. On a stable regimen of any other anti-Parkinson's drugs for at least four weeks before randomization.
9. Be at least 20 years of age.
10. Be willing and able to give written informed consent.

Exclusion Criteria:

1. Taking any excluded medications.
2. Neurosurgical treatment or Transcranial Magnetic Stimulation for PD.
3. Diagnosis of cancer within 5 years.
4. Diagnosis of clinically significant illness of any organ system.
5. Diagnosis of dementia or mini-mental status examination score of 25 or less.
6. History of drug or alcohol abuse or dependence within the past two years.
7. History of psychosis.
8. Significant drug allergies.
9. Taking anticonvulsants for seizures.
10. History of neurological malignant syndrome.
11. Pregnant or lactating females.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the mean total hours of awake time per day spent in the OFF state in patients with Parkinson's disease (PD) treated with levodopa/dopa-decarboxylase inhibitor. | Last Visit

SECONDARY OUTCOMES:
To evaluate the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the mean percentage of awake time per day spent in the OFF state. | Every Visit
To evaluate mean change in the total hours and the percentage of awake time per day spent in the ON state (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia). | Every Visit
To evaluate the change in Unified Parkinson's Disease Rating Scale (UPDRS). | Every Visit
To evaluate change in the Clinical Global Impression - Improvement scale (CGI-I). | Visit 4 and Last Visit
To evaluate the safety of 20 mg/day and 40mg/day doses of istradefylline | Every Visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan